CLINICAL TRIAL: NCT06214299
Title: Study of the Psychometric Properties of Two Questionnaires for Measuring Disease Flare-up in IBD (Crohn's Disease / Hemorrhagic Rectocolitis)
Brief Title: Study of the Psychometric Properties of Two Questionnaires for Measuring Disease Flare-up in IBD
Acronym: Flare-IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: EPSTEIN Jonathan (Other)
Responsible Party: Sponsor-Investigator, EPSTEIN Jonathan, Doctor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2023PI116
Record Dates: First submitted 2023-12-20; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Chronic Inflammatory Bowel Diseases
Keywords: Psychometric properties; Patient-Reported Outcomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validating two questionnaires for measuring relapse in IBD (Crohn's / UC)

DETAILED DESCRIPTION:
IBD (Chronic Inflammatory Bowel Diseases) includes Crohn's disease and ulcerative colitis (UC). In France, an estimated 300,000 people suffer from IBD (source afa Crohn RCH France).

To our knowledge, there are no Patient Reported Outcomes (PROs) validated in French to measure the relapse phenomenon in IBD. Such an instrument would complement the available indicators and enable clinicians to detect treatment response at an early stage, as well as failure to respond to treatment, as manifested by the resumption or increased frequency of relapses, and thus enable rapid adjustment of the proposed therapeutic strategy.

Two questionnaires have been developed, their psychometric properties need to be studied.

The project's deliverable will therefore be two validated questionnaires for measuring relapse from the patient's perspective in IBD for routine use. For this reason, the questionnaires will be short, simple to use, easy to interpret and designed to integrate online applications for patient self-monitoring of IBD disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient member of the AFA Crohn RCH, and registered in the mailing list
* Person having received full information on the organization of the research and not having objected to his/her participation and to the use of his/her data.

Exclusion Criteria:

- There were no non-inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is all patients who are members of the AFA Crohn RCH and belong to their mailing list.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Structural validity evaluated by a confirmatory factor analysis, thresholds: comparative fit index (CFI)>0.90, Tucker-Lewis index (TLI)>0.90, root mean square error of approximation (RMSEA)<0.08 | day 0
  Psychometric properties measurable in a cross-sectional study as described by the COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN), using classical test theory and item response theory

SECONDARY OUTCOMES:
Reproducibility evaluated by answers to respondents' questions according to declared status corresponding to current absence of relapse. Measured by intraclass correlation coefficient (ICC), a value above 0.70 is expected for acceptable reproducibility | day 15
  Reproductibility

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricci L, Toussaint Y, Becker J, Najjar H, Renier A, Choukour M, Buisson A, Devos C, Epstein J, Peyrin Biroulet L, Guillemin F. Web-based and machine learning approaches for identification of patient-reported outcomes in inflammatory bowel disease. Dig Liver Dis. 2022 Apr;54(4):483-489. doi: 10.1016/j.dld.2021.09.005. Epub 2021 Sep 26. PMID 34588153
- See also: Web-based and machine learning approaches for identification of patient-reported outcomes in inflammatory bowel disease — https://pubmed.ncbi.nlm.nih.gov/34588153/